CLINICAL TRIAL: NCT00886002
Title: Explorative, Double-blind Study on Dose Effectiveness of DUROGESIC D-Trans 12 Mcg/h and 25mcg/h Compared to Transtec and Placebo in Acute Pain Models in Healthy Volunteers.
Brief Title: Comparison of Two Dosage Strengths of Transdermal Fentanyl Versus Transdermal Buprenorphine and Placebo in Acute Pain Models in Healthy Volunteers.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen-Cilag A.G., Switzerland (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CR002443
Record Dates: First submitted 2009-04-20; First posted 2009-04-22 (Estimated); Last update posted 2010-06-22 (Estimated); Status verified 2010-06

CONDITIONS: Pain
Keywords: Healthy volunteers
MeSH Terms: conditions — Pain | interventions — Fentanyl; Buprenorphine; Naloxone

INTERVENTIONS:
Drug: Fentanyl; Buprenorphine; Naloxone

SUMMARY:
The primary objective of this pilot trial is to identify pain model(s) which allow(s) to compare and differentiate the analgesic effects between transdermal fentanyl 25Âµg/h, transdermal fentanyl 12Âµg/h and placebo in a dose dependent way. The second objective is to compare the effects of transdermal buprenorphine 35Âµg/h in these models with the effect of the two transdermal fentanyl dosages. Therefore four different treatments are given; all treatments will be by means of a patch that is attached to the back for 72 hours.

DETAILED DESCRIPTION:
After having read and signed the written informed consent form, patients will participate in a screening visit (within 2 weeks before study start, see above selection of study participants). Patients will participate in a training session to experience the three pain test procedures and to assure whether they are able to perform the tests and they are willing to accept these stimuli during the study. They will be hospitalized for 4 treatment cycles (4 days / 5 nights each during which the 4 treatments mentioned under 'Purpose of the Study' are given). Between the hospitalizations they are not required to come to us. The new day -1 for the next cycle is at the same day of the week 2 weeks after the previous hospitalization. For each treatment cycle they enter the facility in the evening (day -1) before the patch is administered and may leave in the morning of day 5. Assessments will be made as follows:

Evening of Day -1: urine drug and alcohol screen, pregnancy test for females, interview by the study physician in charge Days 1, 2, 3, 4, and 5 in the morning: vital signs, pulsoximetry (assessment of oxygen saturation by means of a finger clip) From Day 1 in the morning to Day 5 in the morning: continuous ECG From Day 1 in the morning to Day 4 in the morning: patch administration on the back Days 1, 2, and 4 in the morning: three pain tests*, pupillometry (measurement of the pupil size by a photographic device), blood sample for the measurement of the drug plasma concentrations prior to patch administration in the morning of day 1 they perform three pain tests* (heat, cold pressure test, electric stimulation at the forearm) to assess baseline values and the skin will be checked at the designated patch locations. Patch adhesion will be checked regularly after administration. Patients will be asked regularly during your stay in the unit about concomitant medications and whether any adverse event occurred. In the morning of day 5, before dismission, a physical exam will be performed. The skin underneath the patch will be assessed after removal. After the fourth hospitalisation phase they will leave the facility and they have to return for an ambulant follow up visit 6 - 9 days thereafter. Vital signs will be recorded, they will be asked about concomitant medications and adverse events, a physical exam, clinical laboratory, vital signs and an electrocardiogram will be performed. After this visit the study is terminated. The electrical stimulation model uses a commercially available and registered for human use constant current device delivering wave pulses of 3-s duration. Two electrodes are applied to the lateral lower arm. To determine pain threshold an ascending staircase design is used starting with randomly varied stimuli. The intensity of the stimulus is increased until the pain threshold is reached and afterwards further increased until the maximally tolerated pain is reached. Once pain threshold and the maximally tolerated stimulus are identified, a series of stimuli evenly spaced between a stimulus 30% less than the pain threshold and the maximally tolerated stimulus is administered in a random fashion and the patient rates the pain on a visual analogue scale (VAS).

Heat test: A thermode will be applied on the forearm. The temperature of the thermode will be continuously increased from 30 C to a maximum of 56 C. They will be asked to give a signal when perceiving the heat as painful and to press the bottom when feeling the heat as intolerable pain and not wanting the heat to be further increased.

Cold pressor test: The left hand will be immersed in ice-saturated water for a maximum of 2 min. If pain is felt as intolerable before 2 min have elapsed, they can withdraw the hand. Perceived pain intensity will be rated continuously on a 10 mm visual analogue scale and recorded. Patients will receive one of four treatments one after another: transdermal fentanyl 25 mcg/h, transdermal fentanyl 12 mcg/h, transdermal buprenorphine 35 mcg/h,placebo. All of these treatments are administered as patches. Treatment duration per patch is 72 hours. After this time the patch is removed. Before the next patch of the following treatment will be applied, there will be 11 days without any drug administration. Total duration of the study is 56 days.

ELIGIBILITY:
Inclusion Criteria:

* Healthy on the basis of a pre-study physical examination
* Subjects who are willing to be hospitalized
* subjects who are willing and able to participate in the pain tests and show responsive pain pattern

Exclusion Criteria:

* History or presence of liver or renal insufficiency
* acute liver inflammation, significant cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, haematologic, psychiatric or metabolic disturbances
* severe restriction of respiratory function
* treatment with MAO inhibitors during the last four weeks
* active skin disease or skin irritation at designated patch locations
* history of chronic pain (episodes of more than three months of chronic pain)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2004-11; Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
The first objective of the trial is to identify which acute pain model differentiates best between placebo and transdermal fentanyl 25µg/h.

SECONDARY OUTCOMES:
The second objective is to investigate, whether a significant dosage effect correlation exists in the target model between transdermal fentanyl 25µg/h, 12µg/h and placebo and TRANSTEC 35 mcg/h.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag A.G. Clinical Trial, Study Director — Janssen-Cilag A.G.